CLINICAL TRIAL: NCT02562638
Title: Do Patients Need Pre-Procedural Fasting for Coronary Artery Procedures?
Brief Title: Pre-Procedural Fasting in Cardiac Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-8178-A
Record Dates: First submitted 2015-09-14; First posted 2015-09-29 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Fasting
Keywords: NPO; NBM; pre-procedure; cardiac
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 Fasting (No Intervention): Group 1(control group) Fasting for both solids and fluids for up to 4 hours pre-procedure
- Group 2 Non-fasting (Experimental): Group 2 (intervention arm) Clear fluids up to 1 hour before the procedure and fasting for solids up to 4 hours pre-procedure
  Interventions: Other: Non-fasting

INTERVENTIONS:
Other: Non-fasting — Clear fluids up to 1hour pre-procedure and fasting for solids for up to 4 hours
  Arms: Group 2 Non-fasting

SUMMARY:
Traditionally, patients are kept nil-per-os (NPO) or nil-by-mouth (NBM) prior to invasive cardiac procedures. There exists neither clear evidence nor guidance about the benefits of this.

The investigators aim to assess if there is a reduced incidence of vasovagal complications (primary outcome) and the combined incidence of aspiration pneumonia, change in eGFR, participant satisfaction if participants are not kept fasting.

This (pilot) randomised control trial will have an intervention arm allowing participants to drink clear liquids freely up to 1 hour before the procedure versus keeping them traditionally NPO.

240 patients will be randomised with 120 participants in each arm.

DETAILED DESCRIPTION:
Introduction, background and justification for the study

Patients are traditionally kept Nulla-Per-Os/Nil-By-Mouth (NPO/NBM) for 4-6 hours prior to cardiac procedures including: diagnostic coronary angiograms, right heart catheters, percutaneous coronary interventions and device therapies to minimize the risk of vomiting and pulmonary aspiration during sedation or general anesthesia. The risk of developing pulmonary aspiration is 0.0015 % following emergency coronary artery bypass (CABG) surgery in patients without pre-procedural fasting. There is currently no data available regarding the risk of aspiration during cardiac angiographic interventions, but the risk is likely lower than that of emergency CABG. Currently no North-American or European guidelines require patients to be fasted before cardiac procedures.

The incidence of emergency CABG following cardiac catheterization is between 0.15 % to 0.4 %, whilst that of cardiac arrest is about 1%. In the subset of patients who develop cardiac arrest during elective cardiac catheterization or PCI, the incidence of pulmonary aspiration is low and similar between survivors and non-survivors (8.9% of patients who developed cardiac arrest).

Unsurprisingly, patients admitted with acute MI undergoing Primary PCI (PPCI) are not fasted beforehand and the need for emergency intubation/CABG remains rare in these patients.

A study has shown a rare occurrence of pulmonary aspiration in general anesthesia with a risk of 0.02% for elective and 0.1% for emergency procedures. In two randomized controlled trials, no case of pulmonary aspiration was reported despite the absence of pre-procedure fasting and use of Midazolam/Diazepam/etomidate.

Similarly, in an observational study no patient developed pulmonary aspiration. A Cochrane review did not show an increased risk of pulmonary aspiration with shorter fluid fast. A review article did not report an increased risk of pulmonary aspiration in non-fasted patients in the emergency department. However, a prospective multicenter emergency-department study of 2623 patients revealed only one patient developed aspiration pneumonia following the use of sedation. There is current consensus in the anesthesia literature that it is safe for healthy individuals to drink clear fluids up to 2 hours before induction of general anesthesia. It is recommended that 2 hours fasting for clear fluids, 6 hours for solids and supports the concept of pre-operative oral nutrition using a special carbohydrate-rich beverage. On the other hand, coronary procedures require the use of intravenous contrast, which can precipitate acute renal impairment. It has been shown that proper hydration can reduce the risk of contrast-induced nephropathy. A review study suggests that the oral route is as effective as the intravenous route for volume expansion and reduction of contrast-induced acute kidney injury. A prospective study demonstrated that lack of fasting was not associated with a higher incidence of adverse events in children undergoing pre-procedural sedation in the emergency department. A recent clinical policy published by the American College of Emergency Physicians; has recommended (Level B), that procedural sedations in emergency departments should not be delayed based on fasting status.

Similarly, a recent retrospective study of 1900 patients in UK, demonstrated that patients do not need to be NPO prior to Percutaneous Coronary Intervention (PCI). Another study has demonstrated that reduced gastric pH (<2.0) and increased gastric volumes predisposed to pulmonary aspiration. Invasive procedures such as angiography and angioplasty both are associated with a small risk of adverse events. One such adverse event is vasovagal reaction which occurs in 3-4% of patients and may be exacerbated by depletion of volume as seen in the fasted state .

Current status at the University Health Network UHN policy requires patients to fast for both solids and liquids for a minimum of 4 hours before cardiac catheterization.

The investigators explore a fasting protocol that is different from current UHN policy

Introduction, background and justification for the study:

UHN policy requires patients to fast for both solids and liquids for a minimum of 4 hours before cardiac catheterization.

The investigators explore a fasting protocol that is different from current UHN policy and have involved staff from both the cardiothoracic surgery and anesthesiology teams, who will also act as a safety monitor and be part of the Data Safety Monitoring Board to ensure that participants are safe from harm or adverse effects.

Currently there is no published data on the association between fasting state and peri-procedural vasovagal symptom reduction or procedural satisfaction.

Hypothesis:

A more liberal fasting protocol (fasting > 4 hours for solid, but encouraging oral clear fluids up to 1 hour prior to the procedure) is associated with a lower incidence of peri-procedural vasovagal complications than current standard fasting protocol (> 4 hours for both solids and fluids)

Methods and experimental design:

This is a prospective single-blind randomized pilot study. The Cardiac Interventionists involved in the procedure will be blinded to randomization. All patients undergoing cardiac invasive procedures will be screened for eligibility. The participants will be randomised to 2 groups (eligibility criteria and outcome measures are mentioned in a different section).

Study Groups Group 1 - Control Group: Participants will be fasted according to current standard practice at UHN (a minimum of 4 hours of fasting period for both liquids and solid food).

Group 2 - Intervention group: Participants will be allowed (and encouraged) to drink clear fluids up to 1 hour before the procedure. Solid foods will be allowed up to 4 hours before the procedure which is current standard practice at UHN.

Enrolment and randomization:

Participants who qualify for the study will be approached in person prior to (if in-patient) or on the day of the procedure (if ambulatory) to obtain written informed consent prior to randomization.

A verbal explanation and written information in the form of the patient information sheet will be given to participants. They will be approached by co-investigators who are not involved in their care and given at least 4-24 hours to consent for the study. They will have as much time as they need to consider the study. They will also have the opportunity to discuss it with their family, friends and family doctor.

They will be given contact details of the on-site research team including the study doctors and nurses who will be able to answer any of their queries at any point during the study. They will be notified that they are not obliged to participate in the study and if they do decide to take part and change their mind at any point they can withdraw from the study unconditionally and their withdrawal will not affect their future care.

Vulnerable groups will not be participating in this research hence no special measures will be taken for their recruitment. Participants will also be informed of any potential safety concern that may arise during the study and will be advised about further treatment options. Wherever possible the Hospitals translation service will be used to offer translation of the consent form to patients who do not have English as their first language. Other individuals, who require specialist communication such as the visually impaired or those who suffer from deafness will wherever possible, be accommodated with the hospitals on-site services.

Throughout the study the participant's identity will be protected and will not be disclosed outside the Hospital in keeping with the University Hospital Network (UHN) Patient Health Information (PHI) policy. At the beginning of the study the investigators will receive an identification log to enable them to record patient study pseudonymised identification numbers. This record will remain at the central research offices at the participating centers and will act as a reference document for the PI. Data from the case report forms (CRFs) will be stored on an onsite computer. The hard copy CRFs will be kept in the research doctor's office -the persons able to access the case report forms will be the PI and the cardiology research doctors and nurses delegated for this study purpose.

Follow up:

Participants will be requested to return for one blood test between day 3 and day 5 post- procedure. To and from public transport cost will be provided to the patient and one accompanying person if needed. A telephonic follow up will also be undertaken at one week to ensure no adverse events have occurred.

Baseline investigations/Information:

At the time of the procedure , the investigators will obtain and record the following:

Pre-procedural Information

1. Pre-procedure investigations (Hemoglobin, Urea, Creatinine, eGFR)
2. Patient demographics (Diabetes Mellitus {DM}, hypertension {HTN}, renal impairment, peripheral vascular disease {PVD})
3. Index admission diagnosis (NSTEMI, Chronic stable angina)
4. Weight, height and Body Mass Index (BMI)
5. Medications on admission

Procedural and post-procedural information will be recorded, including:

1. Type of procedure
2. Route (access site-femoral or radial) of procedure
3. Intra-procedural details (sedation, analgesia, complications, devices-used)
4. Procedural and post-procedural outcomes(Success, in-hospital complications, discharge time and date, complications including mortality and aspiration pneumonia)
5. Patient satisfaction survey
6. Post-procedural creatinine
7. Post-procedural telephonic call one week from date of procedure Statistical analysis Demographic and procedural variables will be presented as percentage (categorical variable) or mean ± SD (continuous variable). Comparison of demographic and procedural variables between the two groups will be performed by chi-square or Fisher's exact test for categorical variables and student's t test for continuous variables. Statistical analysis will be performed using SPSS version 22. Randomization will be performed by systematic random sampling by utilizing an online computer generated random number assignment tool.

Sample size calculation:

Sample size was calculated based on proportion and effect size. A total sample size of 240 patients (120 patients in each arm) would have an 80 % power to detect a 1.0% incidence of vasovagal reaction in the intervention arm (for an α of 0.05).

Funding:

This study is being funded by the UHN Innovation Committee. Once the outcomes of the pilot study are available and if safety endpoints are accomplished, , the investigators will consider conducting a similar multicentre study.

Ethics:

All aspects of Good Clinical Practice will be adhered to. Patient confidentiality will be maintained as per the data protection policy including anonymising data. Ethical approval has been obtained from the REB through routine channels (CAPCR).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent
2. Diagnostic coronary angiography and coronary interventions (both elective and stable Acute Coronary Syndrome {ACS} patients).
3. ≥ 18 years of age

Exclusion Criteria:

1. Patients who are intubated
2. Patients unable to give informed consent
3. Patients presenting with an acute unstable condition, including:

   1. STEMI
   2. unstable ACS
4. Patients with a history of or at risk for aspiration pneumonia

   * stroke
   * dysphagia
   * severe gastroesophageal reflux disease
5. Patients with known or anticipated difficult airway
6. Patients who request to be allotted to a particular arm of the study
7. Patients who are temporary transfers from other hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary: Reduction in the incidence of vasovagal complications. | 1 day
  The presence of two or more of the following during the cardiac invasive procedure or during sheath removal or while manual pressure is being applied to the site will constitute a positive vasovagal reaction :
  i) Reduced level of consciousness, nausea and vomiting, and cold, clammy, pale skin ii) Reduction in blood pressure to < 100mmHg systolic or > 15% decrease from baseline iii) Reduction in the heart rate to < 60 beats/minute (or if initial heart rate is < 60/minute, a decrease of > 15% from baseline).
  Patients' heart rate and blood pressure will be monitored (continuously) intra-procedure and (every 15 minutes) post-procedure during sheath removal and while manual pressure is being applied. The expected rate of vasovagal reaction in the NPO group is 3% .

SECONDARY OUTCOMES:
Secondary: 1. Patient satisfaction with procedure as assessed by the patient satisfaction survey form. | 1 day
Secondary: 2. Overall incidence of aspiration pneumonia (intra and post-procedural). | 1 week post procedure
Secondary: 3. Post-procedure change serum creatinine (∆creatinine) compared to pre-procedure. | 5 days post procedure
  The difference between a single pre-procedure measurement of serum creatinine and a single post procedure measure of serum creatinine will be calculated as ∆creatinine. The average ∆creatinine in each randomised arm will be compared to assess difference if any.
Secondary: 4. Post-procedure change eGFR (∆eGFR) compared to pre-procedure. | 5 days post procedure
  The difference between a single pre-procedure measurement of eGFR and a single post procedure measure of eGFR will be calculated as ∆eGFR. The average ∆eGFR in each randomised arm will be compared to assess difference if any.
Secondary: 5. Volume of gastric content immediately prior to the cardiac intervention | 1 day
  This will be assessed in a random subset of 60 patients (30 from each Group) by bedside sonography. Using standard portable ultrasound equipment, a bedside gastric examination will be performed by an investigator blinded to group allocation, in a standard manner as previously described . The volume will be measured in millilitres (ml).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, Principal Investigator — University Health Network, Toronto

REFERENCES:
- [Background] Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: a report by the American Society of Anesthesiologist Task Force on Preoperative Fasting. Anesthesiology. 1999 Mar;90(3):896-905. doi: 10.1097/00000542-199903000-00034. No abstract available. PMID 10078693
- [Background] Rosengarten J, Ozkor M, Knight C: Fasting and cardiac catheterization should we be following the evidence; Controversies and consensus in imaging and intervention (C2I2) 2007: V (2); 22-23
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Background] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Background] Williams DO, Holubkov R, Yeh W, Bourassa MG, Al-Bassam M, Block PC, Coady P, Cohen H, Cowley M, Dorros G, Faxon D, Holmes DR, Jacobs A, Kelsey SF, King SB 3rd, Myler R, Slater J, Stanek V, Vlachos HA, Detre KM. Percutaneous coronary intervention in the current era compared with 1985-1986: the National Heart, Lung, and Blood Institute Registries. Circulation. 2000 Dec 12;102(24):2945-51. doi: 10.1161/01.cir.102.24.2945. PMID 11113044
- [Background] Grayson AD, Moore RK, Jackson M, Rathore S, Sastry S, Gray TP, Schofield I, Chauhan A, Ordoubadi FF, Prendergast B, Stables RH; North West Quality Improvement Programme in Cardiac Interventions. Multivariate prediction of major adverse cardiac events after 9914 percutaneous coronary interventions in the north west of England. Heart. 2006 May;92(5):658-63. doi: 10.1136/hrt.2005.066415. Epub 2005 Sep 13. PMID 16159983
- [Background] Webb JG, Solankhi NK, Chugh SK, Amin H, Buller CE, Ricci DR, Humphries K, Penn IM, Carere R. Incidence, correlates, and outcome of cardiac arrest associated with percutaneous coronary intervention. Am J Cardiol. 2002 Dec 1;90(11):1252-4. doi: 10.1016/s0002-9149(02)02846-1. No abstract available. PMID 12450610
- [Background] Nagel EL, Fine EG, Krischer JP, Davis JH. Complications of CPR. Crit Care Med. 1981 May;9(5):424. doi: 10.1097/00003246-198105000-00037. No abstract available. PMID 7214982
- [Background] Wharton TP Jr. Should patients with acute myocardial infraction be transferred to a tertiary center for primary angioplasty or receive it at qualified hospitals in community? The case for community hospital angioplasty. Circulation. 2005 Nov 29;112(22):3509-20; discussion 3534. doi: 10.1161/CIRCULATIONAHA.104.478362. No abstract available. PMID 16316972
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Wright SW, Chudnofsky CR, Dronen SC, Kothari R, Birrer P, Blanton DM, Bruner A. Comparison of midazolam and diazepam for conscious sedation in the emergency department. Ann Emerg Med. 1993 Feb;22(2):201-5. doi: 10.1016/s0196-0644(05)80203-3. PMID 8427432
- [Background] Chan KLL. Etomidate and midazolam for procedural sedation in the emergency department of Queen Elizabeth Hospital: a randomised controlled trial. Hong Kong J Emerg Med 2008; 15: 75-87.
- [Background] Dunn T, Mossop D, Newton A, Gammon A. Propofol for procedural sedation in the emergency department. Emerg Med J. 2007 Jul;24(7):459-61. doi: 10.1136/emj.2007.046714. PMID 17582032
- [Background] Brady M, Kinn S, Stuart P. Preoperative fasting for adults to prevent perioperative complications. Cochrane Database Syst Rev. 2003;(4):CD004423. doi: 10.1002/14651858.CD004423. PMID 14584013
- [Background] Thorpe RJ, Benger J. Pre-procedural fasting in emergency sedation. Emerg Med J. 2010 Apr;27(4):254-61. doi: 10.1136/emj.2008.069120. PMID 20385672
- [Background] Taylor DM, Bell A, Holdgate A, MacBean C, Huynh T, Thom O, Augello M, Millar R, Day R, Williams A, Ritchie P, Pasco J. Risk factors for sedation-related events during procedural sedation in the emergency department. Emerg Med Australas. 2011 Aug;23(4):466-73. doi: 10.1111/j.1742-6723.2011.01419.x. Epub 2011 May 17. PMID 21824314
- [Background] Maltby JR, Sutherland AD, Sale JP, Shaffer EA. Preoperative oral fluids: is a five-hour fast justified prior to elective surgery? Anesth Analg. 1986 Nov;65(11):1112-6. PMID 3767008
- [Background] Phillips S, Hutchinson S, Davidson T. Preoperative drinking does not affect gastric contents. Br J Anaesth. 1993 Jan;70(1):6-9. doi: 10.1093/bja/70.1.6. PMID 8431336
- [Background] Soreide E, Eriksson LI, Hirlekar G, Eriksson H, Henneberg SW, Sandin R, Raeder J; (Task Force on Scandinavian Pre-operative Fasting Guidelines, Clinical Practice Committee Scandinavian Society of Anaesthesiology and Intensive Care Medicine). Pre-operative fasting guidelines: an update. Acta Anaesthesiol Scand. 2005 Sep;49(8):1041-7. doi: 10.1111/j.1399-6576.2005.00781.x. PMID 16095440
- [Background] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Hiremath S, Akbari A, Shabana W, Fergusson DA, Knoll GA. Prevention of contrast-induced acute kidney injury: is simple oral hydration similar to intravenous? A systematic review of the evidence. PLoS One. 2013;8(3):e60009. doi: 10.1371/journal.pone.0060009. Epub 2013 Mar 26. PMID 23555863
- [Background] Agrawal D, Manzi SF, Gupta R, Krauss B. Preprocedural fasting state and adverse events in children undergoing procedural sedation and analgesia in a pediatric emergency department. Ann Emerg Med. 2003 Nov;42(5):636-46. doi: 10.1016/s0196-0644(03)00516-x. PMID 14581915
- [Background] Godwin SA, Burton JH, Gerardo CJ, Hatten BW, Mace SE, Silvers SM, Fesmire FM; American College of Emergency Physicians. Clinical policy: procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2014 Feb;63(2):247-58.e18. doi: 10.1016/j.annemergmed.2013.10.015. PMID 24438649
- [Background] Hamid T, Aleem Q, Lau Y, Singh R, McDonald J, Macdonald JE, Sastry S, Arya S, Bainbridge A, Mudawi T, Balachandran K. Pre-procedural fasting for coronary interventions: is it time to change practice? Heart. 2014 Apr;100(8):658-61. doi: 10.1136/heartjnl-2013-305289. Epub 2014 Feb 12. PMID 24522621
- [Background] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766
- [Background] Dharma S, Shah S, Radadiya R, Vyas C, Pancholy S, Patel T. Nitroglycerin plus diltiazem versus nitroglycerin alone for spasm prophylaxis with transradial approach. J Invasive Cardiol. 2012 Mar;24(3):122-5. PMID 22388304
- [Background] Epstein SE, Stampfer M, Beiser GD. Role of the capacitance and resistance vessels in vasovagal syncope. Circulation. 1968 Apr;37(4):524-33. doi: 10.1161/01.cir.37.4.524. No abstract available. PMID 5649078
- [Background] Sander-Jensen K, Secher NH, Bie P, Warberg J, Schwartz TW. Vagal slowing of the heart during haemorrhage: observations from 20 consecutive hypotensive patients. Br Med J (Clin Res Ed). 1986 Feb 8;292(6517):364-6. doi: 10.1136/bmj.292.6517.364. PMID 3080172
- [Background] S. B. Hulley, S. R. Cummings, W. S. Browner, et al: Designing Clinical Research: Fourth Edition, LWW, 2013.
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Background] Cubillos J, Tse C, Chan VW, Perlas A. Bedside ultrasound assessment of gastric content: an observational study. Can J Anaesth. 2012 Apr;59(4):416-23. doi: 10.1007/s12630-011-9661-9. Epub 2012 Jan 4. PMID 22215523
- [Background] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Background] Kruisselbrink R, Arzola C, Endersby R, Tse C, Chan V, Perlas A. Intra- and interrater reliability of ultrasound assessment of gastric volume. Anesthesiology. 2014 Jul;121(1):46-51. doi: 10.1097/ALN.0000000000000193. PMID 24595113
- See also: Sample size calculation — http://www.sample-size.net/proportions-effect-size/